CLINICAL TRIAL: NCT04670380
Title: Optimizing the Obstetrician's Movement During a Simulated Forceps Operative Vaginal Delivery. A Biomechanical Study Using Optometric Captation (PERFORMAC)
Brief Title: Optimizing the Obstetrician's Movement During a Simulated Forceps Operative Vaginal Delivery (PERFORMAC)
Acronym: PERFORMAC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PERFORMAC
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Obstetric Trauma
MeSH Terms: interventions — Posture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Posture and movement analysis during a simulated forceps vaginal operative delivery — It will be request from each volunteer to perform a vaginal operative delivery using a Suzor's forceps on a mannequin. The condition will be standardized (anterior occiput low fetal presentation). Each participant will be equipped with 34 reflecting markers allowing to record their movement using infra red cameras (VICON system).

SUMMARY:
Operative vaginal delivery is the main risk factor for pelvic floor trauma occurrence and especially for obstetric anal sphincter injuries. These complications are strongly and negatively impact women's health: fecal incontinence, perineal pain, sexual dysfunction.

The risk appears higher in case of operative vaginal delivery assisted by forceps compared to a vacuum delivery. This considered it is likely that optimizing the performance of the operator that perform the operative vaginal delivery will reduce the morbidity associated with this intervention. There are data bout how to optimize the placement of the forceps on the fetal head before performing the delivery but there are no data about the movement of the obstetrician during this intervention.

The objective is to analyse the posture and the movement of the obstetrician during a simulated forceps operative vaginal delivery using a 3D cinematic analysis. Secondary objectives are to analyse the traction force applied on the forceps during the delivery, to describe the different postures in terms of stability and last to compare the self-declared practice to the objectively observed.

This is a prospective study including 40 volunteers (medical doctors and registrars).

Each volunteer will perform a simulated operative vaginal delivery using a Suzor's Forceps on a high fidelity mannequin. Postures and movement will be assessed using optometric analysis. The force of traction will be assessed during the operative delivery thank to a force sensor on the forceps. The self declared practice collected thanks to individual questionnaires will be compared to the observed practice during the simulation.

The prospects are to identify the best posture and movement for performing an operative vaginal delivery and to promote tools for simulation of medical students.

ELIGIBILITY:
Inclusion Criteria:

* Medical doctor or registrar that have an experience of operative vaginal delivery using forceps in their clinical activity

Exclusion Criteria:

* No practice of the forceps at all

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population will be constituted of 40 volunteers that are medical doctor obstetricians or registrar in obstetrics with an experience of the operative vaginal delivery using Suzor's Forceps.
  All the participants will be aged of 18 or more and will give their informed and written free consent before any investigation.
  There is no patient in this study which is a simulation study performed on MD and registrar.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-02 (Estimated)

PRIMARY OUTCOMES:
Analysis of the postures and the movement during the simulated operative vaginal delivery | Day of inclusion
  measures of angles on joints for the different phases of the operative vaginal delivery

SECONDARY OUTCOMES:
Analysis of the traction force during the operative delivery | Day of inclusion
  Continuous measure of the traction force during the delivery (in Newton) thanks to a force sensor implemented in the forceps
Analysis of the postures in terms of stability | Day of inclusion
  Measure of the gravity center projection, the support basis
Compare self-declared practice to the observed practice | Day of inclusion
  Comparison of the postures self-declared in a questionnaire immediately before the simulation to those observed during the simulation

IPD SHARING:
Plan to Share IPD: Undecided